CLINICAL TRIAL: NCT02540824
Title: A Phase II Clinical Trial to Investigate Efficacy and Safety of Apatinib as a Single Agent in RET-fusion Gene Positive Non-small Cell Lung Cancer Who Failed to Previous Treatment.
Brief Title: Study of Apatinib in RET Fusion Positive Advanced Non-small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tongji University (Other)
Responsible Party: Principal Investigator, Caicun Zhou, Professor, Tongji University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FK-1407
Record Dates: First submitted 2015-08-29; First posted 2015-09-04 (Estimated); Last update posted 2015-09-04 (Estimated); Status verified 2015-09

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Apatinib; RET; gene fusion; Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Apatinib single agent arm (Experimental): Apatinib, single agent, 750mg once daily p.o until disease progression
  Interventions: Drug: Apatinib single agent arm

INTERVENTIONS:
Drug: Apatinib single agent arm — For RET-fusion positive advanced NSCLC patients who failed to previous treatment,treat with apatinib, single agent, 750mg once daily, p.o until disease progression
  Other Names: YN968D1

SUMMARY:
RET fusions are present in 1% to 2% of unselected population of non-small cell lung cancer (NSCLC). Existing US Food and Drug Administration-approved inhibitors of RET tyrosine kinase show promising therapeutic effects in a non-small cell lung cancer patients. Apatinib is an oral multi-kinase inhibitors including RET fusions. This study is designed to evaluate the safety and tolerability of Apatinib in patients with RET fusion positive advanced NSCLC.

DETAILED DESCRIPTION:
To observe objective response rate (ORR) of apatinib in RET fusion positive pre-treated advanced NSCLC.

To observe Progression free survival （PFS）. To assess the overall survival (OS). To assess safety and tolerability. To evaluate quality of life. To explore the relationship between biomarkers and the toxicity/efficacy of apatinib.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 and ≤80 years.
* ECOG performance status of 0 to 1.
* Life expectancy of more than 12 weeks.
* At least one measurable lesion exists.(RECIST 1.1)
* Histologically or cytologic confirmed RET fusion positive advanced Non-small cell lung cancer who failed to prior therapies.
* Required laboratory values including following parameters: ANC: ≥ 1.5 x 10^9/L, Platelet count: ≥ 80 x 10^9/L, Hemoglobin: ≥ 90 g/L, Total bilirubin: ≤ 1.5 x upper limit of normal, ULN, ALT and AST: ≤ 1.5 x ULN, BUN and creatine clearance rate: ≥ 50 mL/min LVEF: ≥ 50% QTcF: < 470 ms
* Signed informed consent
* Females of child-bearing potential must have negative serum pregnancy test. Sexually active male and those having childbearing potential must practice contraception during the study.

Exclusion Criteria:

* Squamous carcinoma (including adeno-squamous carcinoma), small cell lung cancer
* Subjects with third space fluid that can not be controled by drainage or other methods.
* Obvious cavity or necrosis formed in the tumor
* Uncontrolled hypertension
* Hymoptysis, more than 2.5ml daily
* Thrombosis in 12 months, including pulmonary thrombosis, stroke, or deep venous thrombosis
* Received big surgery, had bone fracture or ulcer in 4 weeks
* Urine protein >++, or urine protein in 24 hours> 1.0g
* pregnant or lactating woman
* Receiving any other antitumor therapy.
* Known history of hypersensitivity to apatinib or any of it components.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | change from baseline in tumor size every 6-8 weeks after the initiation of apatinib, up to 24 months
  To evaluate ORR every 6-8 weeks after initiation of apatinib

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | 24 months
  PFS is evaluated in 24 months since the treatment began
overall survival (OS) | 24 months
  evaluated in the 24th month since the treatment began
Safety and Tolerability as measured by adverse events | 24 months
  Number of Participants with treatment related Adverse Events as Assessed by CTCAE v4.0
quality of life (QOL, measured by questionnaire) | 24 months
  Change from baseline in Pain on the 11 point short pain scale (SPS-11)

CONTACTS AND LOCATIONS:
Overall Officials: Caicun Zhou, MD,PhD, Principal Investigator — Shanghai Pulmonary Hospital, Tongji University
Locations (1):
- Department of Oncology, Shanghai pulmonary hospital, Shanghai, China